CLINICAL TRIAL: NCT04588623
Title: The Effect of Probiotic Modulation of Enteral Dysbiosis on dIsease Activity in Patients With PSoriatic Arthritis
Brief Title: The MEDIPSA Clinical Trial
Acronym: MEDIPSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 32-347 ex 19/20
Record Dates: First submitted 2020-07-27; First posted 2020-10-19 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Psoriatic Arthritis
Keywords: psoriatic arthritis; probiotics; microbiome
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omnibiotic Stress Repair (OBSR) (Active Comparator): After randomisation, patients will receive a box with one sachet containing 3g of OBSR for each day.
  Interventions: Dietary Supplement: Omnibiotic Stress Repair (OBSR)
- Placebo (Placebo Comparator): After randomisation, patients will receive an identical box with one sachet containing 3g of Placebo for each day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Omnibiotic Stress Repair (OBSR) — OBSR is given orally once daily (3g) for 3 months
  Arms: Omnibiotic Stress Repair (OBSR)
Other: Placebo — Placebo is given orally once daily (3g) for 3 months
  Arms: Placebo

SUMMARY:
The main purpose of this study is to validate the positive effect of "Omnibiotic Stress Repair" on patients with active psoriatic Arthritis.

DETAILED DESCRIPTION:
This is a single center, double blind (patients and investigators), Placebo controlled randomized trial.

Consecutive patients with Psoriatic Arthritis (PsA) in moderate disease activity (Psoriatic Arthritis Disease Activity Score: PASDAS >3.2 - <5.4) on a stable treatment (no immunomodulatory treatment change in the last 3 months) with biological (bDMARDs) and/or synthetic disease modifying anti-rheumatic drugs (sDMARDs) and/or glucocorticoids will be included in the study. Clinical assessment will be scheduled at baseline, 12 weeks and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥18 years and <90 years of age
2. PsA according to CASPAR criteria
3. MoDA defined by a PASDAS >3.2 - <5.4
4. Stable immunomodulatory therapy for the last 12 weeks before baseline (no change in bDMARD/sDMARD/glucocorticoid treatment)
5. Written informed consent

Exclusion Criteria:

1. History of bariatric surgery
2. Prior use of probiotics in the last 24 weeks
3. Use of probiotics, other than the study product, during the study period.
4. Antibiotic therapy within the last 4 weeks before inclusion
5. Inflammatory bowel disease
6. Recent (less than 12 weeks) acute myocardial infarction or decompensated heart failure
7. Recent (less than 12 weeks) stroke
8. Known malignancy
9. Inability of the patient to follow the treatment protocol
10. Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Effect on disease activity according to PASDAS categories | 3 months
  To test differences in response according to the Psoriatic Disease Activity Score (PASDAS, range 0-10, higher values indicate higher disease activity) after 3 months of intake of OBSR compared to placebo in PsA patients.
  Difference in response is defined by the different amount of patients shifting from moderate disease activity (PASDAS > 3.2 - < 5.4) to low disease activity or remission (PASDAS ≤ 3.2) in the two groups.

SECONDARY OUTCOMES:
Effect on disease activity according to PASDAS score | 3 and 6 months
  To test differences in disease activity according to the Psoriatic Disease Activity Score (PASDAS, range 0-10, higher values indicate higher disease activity) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Effect on disease activity according to PASDAS categories independent of concomitant medication | 3 months
  To test differences in response according to the Psoriatic Disease Activity Score (PASDAS, range 0-10, higher values indicate higher disease activity) after 3 months of intake of OBSR compared to placebo in PsA patients independent of the concomitant medication. For this analysis a logistic regression analysis will be performed using response as dependent and concomitant medication and OBSR/Placebo as indipendent variables.
Longterm effect on disease activity according to PASDAS categories | 3 and 6 months
  To test differences in response according to the Psoriatic Disease Activity Score (PASDAS, range 0-10, higher values indicate higher disease activity) before and after probiotic intake at 3 and 6 months.
  Difference in response is defined by the different amount of patients shifting from moderate disease activity (PASDAS > 3.2 - < 5.4) to low disease activity or remission (PASDAS ≤ 3.2) in the two groups.
Impact of disease according to the PSAID-12 | 3 and 6 months
  To assess differences in disease impact according to the Psoriatic Arthritis Impact of Disease Score - 12 (PSAID-12, range 0-10, higher values indicating worse status) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Impact of disease according to the TJC | 3 and 6 months
  To assess differences in disease impact according to the Tender joint count (TJC, range 0-68, higher values indicating worse status) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Impact of disease according to the SJC | 3 and 6 months
  To assess differences in disease impact according to the Tender joint count (SJC, range 0-66, higher values indicating worse status) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Pain assessed by PtPain VAS | 3 and 6 months
  To assess differences in pain measured by the patient pain visual analogue scale (Pt-VAS, range 0-10, higher values indicating worse status) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Enthesitis assessed by the LEI | 3 and 6 months
  To assess differences in enthesitis according to the leeds enthesitis index (LEI, range 0-6, higher values indicating worse status) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Dactylitis assessed by the DS | 3 and 6 months
  To assess differences in dactylitis according to the dactylitis score (DS, range 0-20, higher values indicating worse status) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Impact of disease according to the PGA | 3 and 6 months
  To assess differences in disease impact according to the Patient global assessment (PGA, range 0-10, higher values indicating worse status) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Impact of disease according to the EGA | 3 and 6 months
  To assess differences in physician's disease assessment according to the Evaluator global assessment (EGA, range 0-10, higher values indicating worse status) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Impact of disease according to the SF-36 | 3 and 6 months
  To assess differences in disease impact according to the Short form health survey 36 (SF-36, Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Dietary assessment according to the Diet-Questionnaire | 3 and 6 months
  To assess differences in diet according to the Diet-Questionnaire (15 questions on the type of diet and amount of food intake. Results will be depicted in a descriptive manner) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Skin involvement according to the PASI | 3 and 6 months
  To assess differences in skin involvement according to the Psoriasis Area and Severity Index (PASI, range 0-72, higher values indicating worse skin involvement) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Impact of skin involvement according to the DLQI | 3 and 6 months
  To assess differences in quality of life due to skin involvement according to the Dermatology Life Quality Index (DLQI, range 0-30, higher values indicating worse quality of life) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Impact of disease according to the HAQ | 3 and 6 months
  To assess differences in disease impact according to the Health Assessment Questionnaire (HAQ, range 0-3, higher values indicating worse status) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Fatigue assessment accoring to the FACIT | 3 and 6 months
  To assess differences in fatigue according to the functional assessment of chronic illness therapy for fatigue (FACIT, range 0-52, higher values indicating worse fatigue) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Hospital anxietey and depression assessment according to the HADS | 3 and 6 months
  To assess differences in hospital anxietey and depression according to the Hospital Anxiety and Depression Scale (HADS, range 0-21, higher values indicating worse status) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Laboratory inflammation assessment according to ESR | 3 and 6 months
  To assess differences in disease impact according to the Erythrocyte sedimentation rate (ESR, mm, higher values indicating worse status) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Laboratory inflammation assessment according to CRP | 3 and 6 months
  To assess differences in laboratory inflammation according to the C-reactive protein (CRP, mg/L. Higher values indicating worse status) before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Change in gut microbiota | 3 and 6 months
  To assess differences in gut microbiota composition (according to 16S rRNA targeted Amplicon Sequencing (%), displayed descriptively) before and after probiotic intake and between the OBSR and placebo control before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Gut permeability according to Zonulin | 3 and 6 months
  To assess differences in gut permeability according to stool Zonulin (ELISA, ng/ml, values above 55 indicate higher permeability) before and after probiotic intake and between the OBSR and placebo control before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Gut inflammation according to Calprotectin | 3 and 6 months
  To assess differences in gut inflammation according to stool Calprotectin (ELISA, mg/l, values above 50 indicate inflammation) before and after probiotic intake and between the OBSR and placebo control before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Neutrophile function according to Phagocytosis assessment | 3 and 6 months
  To assess differences in neutrophile function according to Phagocytosis assessment (Phagotest, normal values 95-99%, lower values indicate less function, Phagoburst, normal values 97-100% (E.coli stimulus), 1-10% (fMLP stimulus), 98-100% (PMA stimulus) before and after probiotic intake and between the OBSR and placebo control before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Inflammation assessment according to cytokine Level | 3 and 6 months
  To assess differences in cytokine levels in blood and synovial fluid (Interleukin (IL) pg/ml with normal ranges: IL-1 (<238), IL-5 (<19.27), IL-6 (<7.0), IL-8 (<10.59), IL-10 (<10.05), IL-17A (<11.14), IL-18 (37.43), IFN Alpha (<1.80), IFN Gamma (<6.82), TNF Alpha (<18.88)) before and after probiotic intake and between the OBSR and placebo control before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Lymphocyte subtypes according to FACS | 3 and 6 months
  To assess differences in lymphocyte subtypes according to fluorescence activated cell sorting (FACS, %) before and after probiotic intake and between the OBSR and placebo control before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.
Metabolic assessment using NMR | 3 and 6 months
  To assess metabolomic differences in stool, serum and synovial fluid using nuclear magnetic resonance (NMR metabolic profiling, results are shown in a descriptive manner) before and after probiotic intake and between the OBSR and placebo control before and after probiotic intake at 3 and 6 months and between the OBSR and placebo control group at 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No